CLINICAL TRIAL: NCT06250738
Title: Shift-and-persist and Cardiometabolic Markers Among Women in Puerto Rico: A Pilot of a Mindfulness-based Trial
Brief Title: Shift-and-persist and Cardiometabolic Markers Among Women in Puerto Rico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Andrea Lopez-Cepero, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006752; 8K12AR084234 (NIH)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Psychological Distress; Cardiometabolic Syndrome
Keywords: Mindfulness-based Stress reduction programs; Cardiometabolic outcomes; Psychological well-being; Health behaviors
MeSH Terms: conditions — Metabolic Syndrome; Psychological Well-Being; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental)
  Interventions: Behavioral: Mindfulness-based Stress reduction program: Virtual; Behavioral: Home exercises

INTERVENTIONS:
Behavioral: Mindfulness-based Stress reduction program: Virtual — Through mindfulness meditation and a series of carefully crafted exercises, MBSR equips individuals with powerful tools to manage stress, reduce anxiety, and enhance their overall well-being. Participants will complete 4 weekly virtual sessions covering topics like introduction to stress and its consequences, awareness of sensations, and thoughts, mindful eating, and mindful walking.
Behavioral: Home exercises — Following each virtual session, participants will be given home exercises like practicing awareness of breathing, awareness of thoughts, and awareness of eating.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of a 4-week mindfulness program among young women in Puerto Rico with elevated stress. The main questions it aims to answer are:

* how feasible and acceptable is a s a 4-week mindfulness program among participants with elevated stress
* what are the changes in psychological resilience, psychological distress, health behaviors, and cardiometabolic markers

Participants will be asked to

* attend 4 weekly virtual sessions and daily mindfulness exercises at home
* complete online study questionnaires

DETAILED DESCRIPTION:
Cardiometabolic diseases among women in Puerto Rico. The 1.7 million women residing in Puerto Rico experience a great load of cardiometabolic diseases (i.e., adiposity, type 2 diabetes, hypertension, and hyperlipidemia). It is estimated that, among women in PR, the prevalence of overweight and obesity is 67.1%, hypertension 39.2%, hyperlipidemia 36.8%, and type 2 diabetes 16.3%, with estimates of obesity and type 2 diabetes being higher than in men. With cardiometabolic diseases driving the majority of deaths and disability in Puerto Rico -including women, the steep societal and individual cost of these diseases-particularly in the context of Puerto Rico's financial crisis, it is imperative to understand modifiable factors influencing women's cardiometabolic health and guide early prevention efforts.

Psychological well-being and cardiometabolic health. Psychological well-being has gained attention as a protective factor against cardiovascular disease. This is of particular importance to women in Puerto Rico as they report greater psychological distress than Puerto Rican men. The protective effect of psychological well-being on cardiometabolic health is believed to partially occur by buffering the effects of stress on health. This is of particular importance to women in Puerto Rico given that stress is detrimental to Latinx cardiometabolic health. Puerto Ricans in the mainland US have lower psychological well-being, as measured by optimism, than other Latinx heritage groups.

Mindfulness-based Stress reduction programs (MBSR). The high burden of cardiometabolic diseases among women in Puerto Rico, their disproportionate exposure to stressors, and potentially low psychological well-being highlight the need for effective behavioral interventions. The American Heart Association has issued a call to action for studies testing mindfulness-based interventions for cardiometabolic health. At its core, this program empowers participants to develop a profound awareness of the present moment, fostering a deeper understanding of their thoughts, emotions, and bodily sensations. Through mindfulness meditation and a series of carefully crafted exercises, MBSR equips individuals with powerful tools to manage stress, reduce anxiety, and enhance their overall well-being. MBSR consists of an 8-week program with weekly sessions (usually lasting 2.5 hours), daily practice exercises (of 45 minutes duration each), and an end-of-program day-long retreat. MBSR has been shown to improve psychological well-being, with studies documenting greater intervention effectiveness and acceptability for women than men. Additionally, studies have shown that mindfulness-based interventions reduce adiposity and hypertension. However, there is limited data on MBSR in Latinx women-less in Puerto Rico. The Puerto Rican population has unique socio-cultural values and norms that merit MBSR to be tested in this group.

MBSR interventions have critical pitfalls, such as time and transportation barriers, that need to be addressed to improve implementation. The only study in Puerto Rico evaluating an MBSR reported time commitment and lack of transportation as barriers to participation. A study done at UMass Medical School did some preliminary work to address these limitations. The researchers at UMass have adapted the original MBSR to use shortened weekly sessions (1.5- 1hr) and home practice exercises (5-15min). The researchers also selected 4 sessions out of the original 8-week MBSR sessions to shorten the program. This responds to preliminary data from our focus group discussions among young women in Puerto Rico documenting that an 8-week long program with weekly sessions was a burden and would hinder participation.

The Investigator took these modifications and further made adaptations to make the 4-week MBSR program be delivered virtually. The original 4-week protocol by Rosal and Camrody was already available in English and Spanish. In the present study, we will test the feasibility and acceptability of the Spanish version 4-week MBSR program among young women (18-29yr) with elevated stress residing in Puerto Rico and will explore changes in resilience, stress, health behavior, and cardiometabolic outcomes. Testing the Spanish 4-week MBSR protocol in young women in Puerto Rico is needed to evaluate novel strategies that may be feasible and acceptable for this group

ELIGIBILITY:
Inclusion Criteria:

* Individuals residing in Puerto Rico
* Spanish speaking
* Elevated stress (defined as a score >6 in the Perceived Stress Scale (PSS-4)34)
* Willing to undergo research activities (focus group discussions).

Exclusion Criteria:

* Currently pregnant
* Previous participation in an 8-week MBSR program
* Experiencing moderately severe or severe depressive symptoms (PHQ-9>15)35)
* Have active suicidal ideation (PHQ-9 item #9)35
* Self-report history of cognitive and psychiatric conditions
* Lack of access to the internet/phone (mode of focus group discussions-via Zoom)
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — * Reporting female sex at birth
  * Not identifying as a man, trans man, or trans woman
Enrollment: 24 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lopez-Cepero, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- Rollins School of Public Helath, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on the following variables may be shared: psychological distress (depression symptoms, anxiety symptoms, PTSD symptoms), resilience (shift and persist, mindfulness), health behaviors (smoking, eating habits), weight, blood pressure, height, sociodemographic (socioeconomic variables, age), number of sessions attended and practice exercise completed.
Supporting Information: Study Protocol
Time Frame: 06/2024 - 06/2028
Access Criteria: Investigators interested in conducting analyses will need to submit a manuscript proposal to be reviewed by the PI. Data and study files will be shared upon positive review.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through social media pages and email blasts at academic institutions.
  Participant enrollment began on February 17, 2024, and all 2 months follow-up assessments were completed by April 27, 2024
Period: Overall Study
Arm/Group | Study Population
Started | 24
Completed | 23
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education level [Count of Participants; unit: Participants]
  High school graduate-some college | 6
  Undergraduate | 8
  Graduate | 10
Employment status [Count of Participants; unit: Participants]
  Student | 11
  Working full/part time | 12
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Rates of Recruitment and Retention
Description: Number of participants at the beginning of the study versus the number of participants at the end of the study.
Time Frame: Baseline, week 4, week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 24
Participants
  Baseline | 24
  Week 4 | 24
  Week 8 | 23

2. Primary Outcome: Adherence to the Program: Frequency of Daily Mindfulness Practice Exercises at Home
Description: The frequency of self-reported completed home practice was assessed at post-intervention assessments.
  Participants will answer the question "Usually, how often did you practice the at-home exercises of the program?". Response options include: never, <1/week 1-2/week, 3-4/week, 5-6/week, every day.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 24
Participants
  Never | 0
  < 1/week | 4
  1-2/week | 8
  3-4/week | 8
  5-6/week | 3
  Everyday | 1

3. Primary Outcome: Adherence to the Program: Number of 4-week MBSR Sessions Joined
Description: Measured by the number of sessions joined. This is tracked by session attendance done by research staff". Data entered will be 0 sessions, 1 session, 2 sessions, 3 sessions or 4 sessions
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 24
Participants
  0 sessions | 0
  1 session | 0
  2 sessions | 2
  3 sessions | 2
  4 sessions | 20

4. Primary Outcome: Ratings of Satisfaction (Overall)
Description: Ratings of program satisfaction, also assessed by survey in post-intervention assessments, will be measured with aseveral questions on, including one that reads "Overall, how satisfied were you with the stress reduction program
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 24
Participants
  Very satisfied | 19
  Somewhat satisfied | 4
  Somewhat dissatisfied | 1
  Very Dissatisfied | 0

5. Primary Outcome: Ratings of Satisfaction Pre and Post Intervention
Description: Satisfaction with the ability to manage stress in life before and after the 4-week MBSR intervention
Time Frame: Baseline, week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 24
Participants
  Pre-intervention: Very dissatisfied | 3
  Pre-intervention: Dissatisfied | 16
  Pre-intervention: Satisfied | 4
  Pre-intervention: Very satisfied | 1
  Post-intervention: Very dissatisfied | 0
  Post-intervention: Dissatisfied | 1
  Post-intervention: Satisfied | 6
  Post-intervention: Very satisfied | 17

6. Secondary Outcome: Change in Depression Symptoms: CSED-10 Scores
Description: The CESD-10 is a shortened version of the 20-item CES-D, designed to assess depressive symptoms. It includes 10 questions rated on a 4-point Likert scale (0-3), with higher scores indicating greater symptom severity. The scale covers both negative (e.g., loneliness, sadness) and positive (e.g., hopefulness, happiness) experiences. A total score ranges from 0 to 30, with a score of 10 or higher often indicating significant depressive symptoms and a potential risk for Major Depressive Disorder (MDD).
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 13.4 (5.4)
  Week 4 | 8.3 (6.2)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 8.8 (6.8)

7. Secondary Outcome: Change in Anxiety Symptoms: GAD-7 Scores
Description: The GAD-7 is a seven-item screening tool for generalized anxiety disorder. Each item is rated on a 0-3 scale, with total scores ranging from 0 to 21. Higher scores indicate greater anxiety severity, with 10 or higher suggesting possible GAD. Severity levels range from minimal (0-4) to severe (15-21).
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 9.0 (3.4)
  Week 4 | 6.0 (4.1)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 5.5 (4.6)

8. Secondary Outcome: Change in PTSD Symptoms: Civilian Abbreviated Scale
Description: Two symptoms of PTSD experienced in the previous month were assessed with the PTSD Civilian Abbreviated Scale. One item measured disturbing memories of any adverse event, and the second item measured feelings of distress due to these memories.
  Response options to both items were on a 5-point scale and ranged from 0 'not at all' to 4 'extremely'. Response options to both items were summed (Lowest score: 0, highest score: 8), with higher scores indicating greater PTSD symptomatology.
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 6.6 (2.0)
  Week 4 | 4.8 (1.6)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 4.3 (1.6)

9. Secondary Outcome: Change in Perceived Stress (Perceived Stress Scale)
Description: The PSS-4 is a short tool measuring perceived stress based on feelings of unpredictability and overwhelm. Scores range from 0 to 16, with higher scores indicating greater stress.
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 8.7 (1.9)
  Week 4 | 6.0 (3.0)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 5.7 (3.1)

10. Secondary Outcome: Shift-and-persist (Chen et al)
Description: It includes 8 items: 4 measuring shift and 4 measuring persist. Response options for all items were on a 4-point Likert scale (from a score of 1 for 'not at all' to a score of 4 for 'a lot'). Total scores were calculated by summing each subscale's items, and possible scores range from 8 to 32, with higher scores indicating greater shift and persist
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 24.0 (4.7)
  Week 4 | 26.5 (4.9)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 26.6 (4.7)

11. Secondary Outcome: Change in Mindfulness: Five Facet Mindfulness Questionnaire (FFMQ-15)
Description: The FFMQ-15 is a 15-item tool assessing mindfulness across five dimensions: observing, describing, awareness, non-judging, and non-reacting. Higher scores indicate greater mindfulness, linked to better emotional regulation and well-being.
  Average scores are obtained by adding up the responses and dividing by the total number of items, reflecting the overall agreement with each item (1 = rarely true, 5 = always true). Higher scores suggest a greater level of mindfulness in daily life.
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 3.1 (0.5)
  Week 4 | 3.4 (0.6)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 3.5 (0.7)

12. Secondary Outcome: Change in Psychological Flexibility: Acceptance and Action Questionnaire - II
Description: The AAQ-II measures psychological flexibility, or the ability to accept negative emotions and take value-driven actions. Higher scores indicate greater flexibility, associated with better emotional resilience and well-being.
  Includes seven statements that participants rate using a 7-point Likert scale, from 1 ("Never true") to 7 ("Always true"). The total score is obtained by adding the ratings for all items (ranging from 7- 49). Higher scores reflect lower psychological flexibility, whereas lower scores indicate greater flexibility
Time Frame: Baseline, week 4, 2 month follow up
Population: 1 subject was lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 24
score on a scale
  Baseline | 24.0 (9.5)
  Week 4 | 17.9 (8.9)
  2 month Follow up: number analyzed (Participants) | 23
  2 month Follow up | 18.1 (10.1)

ADVERSE EVENTS:
Time Frame: Starting from baseline until 2 month follow-up.
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT06250738/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT06250738/ICF_000.pdf